CLINICAL TRIAL: NCT01468662
Title: Cardiovascular Magnetic Resonance Scan Repeatability in ST Segment Elevation Myocardial Infarction
Brief Title: CMR Repeatability in STEMI
Status: Completed | Type: Observational
Sponsor: University of Bristol (Other)
Responsible Party: Principal Investigator, Elisa McAlindon, Cardiology Clinical Research Fellow, University of Bristol
Other Study IDs: Study 1569
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI

SUMMARY:
The investigators propose to conduct a study to measure the reproducibility of CMR parameters that have been used to predict outcome following PPCI: infarct size, left ventricular volumes, myocardial salvage, microvascular obstruction (MVO) and myocardial oedema.

ELIGIBILITY:
Inclusion Criteria:

Participant may enter study if ALL of the following apply

1. ST segment myocardial infarction as defined by ECG (by 2 contiguous limb leads with >1 mm ST-segment elevation, or >2 mm ST-segment elevation in contiguous precordial leads, or new LBBB) and > 20 minutes of cardiac chest pain
2. Written informed consent

Exclusion Criteria:

Participant may not enter study if ANY of the following apply

1. Contraindication to MRI (implanted pacemaker/ defibrillator, ferromagnetic metal implant/ injury, claustrophobia, obesity/ too large for CMR scanner)
2. Known allergy to gadolinium
3. Chronic atrial fibrillation
4. Renal impairment with eGFR <30
5. Cardiogenic shock
6. Patients with special communication needs

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ST segment elevation myocardial infarction
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Inter-observer, intra-observer and inter-scan variability and agreement | Between 2 scans

CONTACTS AND LOCATIONS:
Overall Officials: Elisa McAlindon, BMBS, Principal Investigator — University of Bristol
Locations (1):
- Bristol Heart Institute, Bristol, United Kingdom

REFERENCES:
- [Derived] McAlindon EJ, Pufulete M, Harris JM, Lawton CB, Moon JC, Manghat N, Hamilton MC, Weale PJ, Bucciarelli-Ducci C. Measurement of myocardium at risk with cardiovascular MR: comparison of techniques for edema imaging. Radiology. 2015 Apr;275(1):61-70. doi: 10.1148/radiol.14131980. Epub 2014 Oct 21. PMID 25333474